CLINICAL TRIAL: NCT00371995
Title: The Efficacy and Safety of a Short Course of Miltefosine and Liposomal Amphotericin B for Visceral Leishmaniasis in India
Brief Title: Short Course of Miltefosine and Liposomal Amphotericin B for Kala-azar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Collaborators: Rajendra Memorial Research Institute of Medical Sciences (Other)
Responsible Party: Shyam Sundar, Professor, Banaras Hdindu University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEI PDE 06 03
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2008-09

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; kala-azar; miltefosine; AmBisome
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B; miltefosine

ARMS (1):
- 1 (Experimental): Liposomal amphotericin B administered intravenously as single dose on day 1, Dosage: 5 mg/kg.
  Miltefosine administered orally (50 mg capsules) for 14 days (on days 2-15)
  Interventions: Drug: Liposomal amphotericin B and Miltefosine

INTERVENTIONS:
Drug: Liposomal amphotericin B and Miltefosine — Liposomal amphotericin B administered intravenously as single dose on day 1, Dosage: 5 mg/kg.
  Miltefosine administered orally (50 mg capsules) for 14 days (on days 2-15)
  Other Names: AmBisome and Impavido

SUMMARY:
Miltefosine and liposomal amphotericin B (AmBisome) are approved drugs for visceral leishmaniasis. In this study both drugs will be given in a sequential manner. AmBisome will be given on day 1, followed by Miltefosine for 14 days. Final Cure will be evaluated at six months.

DETAILED DESCRIPTION:
Methodology Multicenter trial, eligible patients will be treated with Liposomal amphotericin B (5 mg/kg) on day 1 and then with miltefosine capsules for 14 days (days 2-15).

At two weeks after the end of treatment the initial cure (clinical and parasitological cure) and the clinical response will be determined. If initial cure is observed, a patient will be evaluated after a 6 months (after end of treatment) follow up period for final clinical cure.

Number of patients planned Total number of patients planned: 150 patients at both centers combined. 75 pediatric (2-11 years); 75 adult (12-65 years).

Lack of suitability for the trial:

* Post Kala-azar Dermal Leishmaniasis (PKDL)
* Concomitant treatment with other anti-leishmanial drugs
* Any condition which compromises ability to comply with the study procedures

Administrative reasons:

* Any condition or situation that compromises compliance with study procedures including follow-up visit Study medication, dose and mode of administration Liposomal amphotericin B administered intravenously as single dose on day 1, Dosage: 5 mg/kg.

Miltefosine administered orally (50 mg capsules) for 14 days (on days 2-15)

Dosage:

1. weighing ≥ 25 kg: 100 mg miltefosine daily as one capsule (50 mg) in the morning and one capsule in the evening, after meals for 14 days.
2. weighing < 25 kg: 50 mg miltefosine daily as one capsule (50 mg) in the morning, after meals for 14 days. Parameter for evaluation

   * Final cure rate (initial parasite cure and clinical assessment at six month EOT)
   * Initial parasitological cure rate (based on splenic aspirates or Bone marrow aspirate)
   * Clinical response at end of treatment (clinical assessment)
   * Adverse events

Statistical methods

* Calculation of cure rate with 95% and 90% lower confidence limit according to Clopper Pearson
* Calculation of overall incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Male and female age between 2 and 65 years (inclusive)
* Parasites visualized on splenic aspiration
* Signs and symptoms compatible with visceral leishmaniasis (e.g. fever, splenomegaly, anaemia, weight loss, leucopenia, thrombocytopenia)
* Confirmed diagnosis of VL by visualization of parasites on splenic/bone marrow aspirate
* Fever for at least 2 weeks
* Written informed consent from the patient/or from parent or guardian if under 18 years old

Exclusion Criteria:

* Hemoglobin < 6 g/dl
* White blood cell count < 1000/mm3
* Platelets <50,000
* Prothrombin time > 5 sec above control
* ASAT > 3 times the upper limit of normal
* Serum creatinine or BUN > 1.5 times the upper limit of normal
* Malaria
* Tuberculosis
* HIV positive serology
* Lactation, pregnancy
* Refusing contraception method during treatment period plus 3 months
* Any medical condition(s) that upon judgment of physician may affect the safety of the patient when treated with study drugs
* Any concomitant drug that is nephrotoxic

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Final Cure six months after the end of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Banaras Hindu University; Prabhat K Sinha, MD, Principal Investigator — Rajendra Memorial Research Institute of Medical Sciences
Locations (2):
- India (2):
  - Kala-azar Medical Research Center, Muzaffarpur, Bihar
  - Rajendra Memorial Research Institute of Medical Sciences, Patna, Bihar

REFERENCES:
- [Result] Sundar S, Sinha PK, Verma DK, Kumar N, Alam S, Pandey K, Kumari P, Ravidas V, Chakravarty J, Verma N, Berman J, Ghalib H, Arana B. Ambisome plus miltefosine for Indian patients with kala-azar. Trans R Soc Trop Med Hyg. 2011 Feb;105(2):115-7. doi: 10.1016/j.trstmh.2010.10.008. Epub 2010 Dec 3. PMID 21129762